CLINICAL TRIAL: NCT03462680
Title: GPR109A and Parkinson's Disease: Role of Niacin in Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: N1613-I
Record Dates: First submitted 2018-02-22; First posted 2018-03-12 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Niacin; Niacinamide

STUDY DESIGN:
Intervention Model Description: There are two arms, niacin and placebo. They are double blind and randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only Pharmacists keep the log of the drug dispensed. Everyone else is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- niacin (Active Comparator): Niacin 250 mg is compared to placebo tablet.
  Interventions: Dietary Supplement: niacin
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: niacin — Niacin or nicotinic acid 250 mg tablets
  Other Names: vitamin B3
  Arms: niacin
Other: placebo — placebo tablet
  Arms: placebo

SUMMARY:
Inflammation plays a central role in Parkinson's disease. The use of anti-inflammatory drugs was found to reduce the risk of PD . Niacin may play an important role in reducing inflammation in PD. The investigators also found that individuals with PD have a chronic niacin deficiency .

The purposes of this study are to (1) examine the blood, urine and spinal fluid of persons with Parkinson's to look for evidence of inflammation and; (2) whether 6 months of vitamin B3 supplements may reduce the inflammation and/or improve symptoms.

DETAILED DESCRIPTION:
Inflammation plays a central role in Parkinson's disease (PD) pathology [1] as evidenced by the presence of microglia in the substantia nigra in post-mortem samples [2] as well as activated microglia and cytokines in clinical and animal studies [3]. The use of non-aspirin non-steroidal anti-inflammatory drugs was found to reduce the risk of PD [4]. The investigators recently identified an anti-inflammatory receptor GPR109A that is upregulated in PD [5]. Niacin has a high affinity for this receptor, suggesting that it (niacin) may play an important role in reducing inflammation in PD. The investigators also found that individuals with PD have a chronic niacin deficiency [5]. Using seed funding from the local PD chapter, the investigators obtained pilot data which suggested that restoring the deficiency via over-the-counter (OTC) supplementation reduced inflammation and decreased the severity of the disease symptoms [6]. In this VA-funded study, the investigators will determine the effect of 6 months' OTC niacin supplementation on inflammation (as assessed in the blood and spinal fluid) and severity of the PD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* PD subjects will be adult men and women diagnosed with idiopathic mild to moderately severe PD defined as modified Hoehn & Yahr Stages I-III (while "On").

  * PD is defined according to the United Kingdom Brain Bank Criteria made at least six months prior to recruitment to the study.
  * PD features include the presence of at least two of the four cardinal clinical manifestations of the disease, which are tremor, rigidity, bradykinesia, and disturbances of posture or gait, without any other known or suspected cause of Parkinsonism.
* Subjects should be stabilized on PD medication for at least 3 months before enrollment into the study.
* Subjects' PD drug prescriptions will not be altered nor withheld during the study, i.e., they will be tested while "On."
* The patient will have signed informed consent.
* Subjects who do not have PD (i.e., healthy or have other medical conditions such as traumatic brain injury (TBI), stroke, or other syndromes in which inflammation plays a role in the condition) will also be recruited as control subjects.
* This will allow us to estimate whether these other conditions show similar or unique inflammatory profile.

Exclusion Criteria:

* Subjects will be excluded if they had previous brain surgery or other severe neurological problems

  * intracerebral hemorrhage
  * traumatic brain injury
  * central nervous system malignancy
  * active central nervous system (CNS) infection
  * significant stroke
  * Alzheimer disease or any type of implanted stimulator including but not limited to Deep Brain Stimulator (DBS) or pacemaker
* All subjects must be without evidence of dementia, defined as a score > 24 the Mini-Mental State Examination and able to understand test instructions
* Subjects must not have functional blindness (inability to participate in gait and visuomotor assessments) or lower limb amputation higher than the forefoot or any orthopedic problem that precludes performance of physical tests
* Allergic to niacin
* Significant cardiac, pulmonary, hepatic, gastrointestinal, or renal disease

  * e.g., New York Heart Association Class III or IV congestive heart failure
  * endocarditis
  * pulmonary insufficiency symptomatic at rest or with mild physical exertion
  * acute or chronic hepatitis
  * renal failure requiring dialysis
  * second and third degree atrioventricular block or sick sinus syndrome), or diabetes are also exclusionary factors

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandramohan Wakade, MBBS, Principal Investigator — Charlie Norwood VA Medical Center, Augusta, GA
Locations (1):
- Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
As the investigators request, we will share the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the study is closed.
Access Criteria: When we are ready to publish, the data will be available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niacin | Placebo
Started | 21 | 26
Completed | 18 | 21
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin | Placebo | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6) | 68 (10.7) | 68.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 19 | 24 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 26 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 23 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 26 | 47
UPDRS III [Mean (Standard Deviation); unit: units on a scale] — The minimum is 0 and the maximum is 120. Higher scores are worse outcomes.
  units on a scale | 21.25 (15.8) | 22.4 (11.8) | 21.9 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Change
Description: This is the Unified Parkinson's disease rating scale assessment. The investigators assess I, II, III and V components of the UPDRS. UPDRS 3 is motor skills. Higher scores mean worse outcome. A 0 is minimum and 120 is the maximum.
Time Frame: at the recruitment and after 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
units on a scale
  baseline | 21.25 (15.8) | 22.4 (11.8)
  6 months | 20.8 (12.4) | 22.31 (16.5)

2. Primary Outcome: REM Sleep Pattern
Description: This requires an instrument Zeo sleep monitor. Subjects are given instructions how to use it. Sleep sensor patches are supposed to be applied on forehead before going to sleep and the data of quality of sleep is captured overnight. The reported data captures the rapid eye movement (REM) sleep as a percentage.
Time Frame: baseline and after 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
percentage of sleep time
  baseline | 20.09 (13.36) | 15.83 (12.1)
  6 months | 21.1 (11.6) | 21.45 (16.3)

3. Primary Outcome: Deep Sleep
Description: This requires an instrument Zeo sleep monitor. Subjects are given instructions how to use it. Sleep sensor patches are supposed to be applied on forehead before going to sleep and the data of quality of sleep is captured overnight. The reported data captures the deep sleep percentage.
Time Frame: At baseline and after 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: percentage of deep sleep time
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
percentage of deep sleep time
  at baseline | 8.17 (5.11) | 8.48 (6.07)
  6 months | 12.28 (16.27) | 8.32 (6.09)

4. Primary Outcome: Light Sleep
Description: This requires an instrument Zeo sleep monitor. Subjects are given instructions how to use it. Sleep sensor patches are supposed to be applied on forehead before going to sleep and the data of quality of sleep is captured overnight. The reported data captures the light sleep percentage.
Time Frame: baseline and 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: percentage of light sleep time
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
percentage of light sleep time
  baseline | 49.2 (17.9) | 53.5 (18.2)
  6 months | 50.9 (15.6) | 47.5 (18.5)

5. Primary Outcome: Sleep Time - Awake
Description: This requires an instrument Zeo sleep monitor. Subjects are given instructions how to use it. Sleep sensor patches are supposed to be applied on forehead before going to sleep and the data of quality of sleep is captured overnight. The reported data captures the awake time during night sleep percentage.
Time Frame: at baseline and 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: percentage of awake-sleep time
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
percentage of awake-sleep time
  baseline | 20.2 (23.23) | 21.95 (17.4)
  6 month | 13.5 (10.3) | 23 (20.7)

6. Primary Outcome: Mini-Mental State Examination (MMSE) Change
Description: It captures mental status and awareness of time, place and surrounding. A zero is minimum and 30 is maximum. Higher score indicates better cognition.
Time Frame: at baseline and after 6 months of treatment
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
score on a scale
  baseline | 29.94 (0.24) | 29.81 (0.88)
  6 months | 29.94 (0.24) | 29.71 (0.78)

7. Primary Outcome: Stroop Test Change
Description: It captures understanding of color and its description within a certain time frame when letters and colors do not match. There are only two choices to pick from and the correct choices should be made to proceed to the next one. Correct choices are given one point and incorrect choices delete one point. Maximum number of correct choices per unit time are recorded. Three initial trials are given to understand the test. No minimum or maximum values. Higher numbers indicate better cognition.
Time Frame: at the baseline and after 6 months of intervention
Population: Stroop test was added after recruitment of few subjects.
Measure: Mean (Standard Deviation); unit: number of correct responses/unit time
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 17
number of correct responses/unit time
  baseline | 6.18 (7.92) | 8.13 (6.64)
  6 months | 8.37 (5.6) | 8.72 (6.86)

8. Primary Outcome: Fatigue Severity Scale
Description: Fatigue was rated from 0-7 in a fatigue questionnaire. A 0 being the least and 7 being the highest level of fatigue.
Time Frame: at baseline and after 6 months
Population: Patients who completed 6 months were analyzed for this measure (39 subjects).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 18 | 21
score on a scale
  baseline | 40.3 (11.99) | 36.7 (13)
  6 months | 38.5 (10.99) | 36.7 (14.2)

9. Secondary Outcome: Cerebrospinal Fluid Changes - Interleukin 6 (IL6)
Description: IL-6 cytokine levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention.
Time Frame: at baseline and after 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 1.6 (0.5) | 1.9 (2)
  6 months | 1.2 (0.37) | 1.2 (0.4)

10. Secondary Outcome: Cerebrospinal Fluid Changes - Interleukin 10 (IL-10)
Description: IL-10 will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention.
Time Frame: at baseline and after 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 0.42 (0.64) | 0.13 (0.16)
  6 months | 0.09 (0.01) | 0.08 (0.04)

11. Secondary Outcome: Niacin Metabolite in Urine - Niacin
Description: Plasma and urine samples will be tested to report levels of niacin and its metabolites. Higher value indicates higher niacin levels
Time Frame: at baseline and after 6 months
Population: A subset of groups were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 23
ng/L
  baseline | 1826.8 (663.2) | 1533 (895.9)
  6 months | 1913.8 (481) | 1660.6 (431.7)

12. Secondary Outcome: Niacin Metabolites in Urine - NAM Nicotinamide
Description: as for outcome 11
Time Frame: at baseline and 6 months
Population: A subset of subjects were randomly selected for this analysis.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 23
ng/L
  baseline | 815.5 (1155) | 205.8 (312.99)
  6 months | 1140.3 (1058.4) | 685.4 (709.3)

13. Secondary Outcome: Niacin Changes in Plasma - Niacin
Description: as for outcome 11
Time Frame: baseline and 6 months
Population: A subset of subjects were randomly selected for this analysis.
Measure: Mean (Standard Deviation); unit: nM/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 22
nM/L
  baseline | 68.5 (95.96) | 55.8 (88.3)
  6 months | 80.83 (92.4) | 92.2 (59.1)

14. Secondary Outcome: Niacin Changes in Plasma - NUA Nicotinuric Acid
Description: as for outcome 11
Time Frame: at baseline and 6 months
Population: Plasma and urine samples will be tested to report levels of niacin and its metabolites. Higher value indicates higher niacin levels. Undetectable values are reported as zero. A subset of the groups were analyzed.
Measure: Mean (Standard Deviation); unit: nM/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 22
nM/L
  at baseline | 0 (0) | 4.99 (17.98)
  6 months | 313.9 (442.7) | 0.38 (1.53)

15. Secondary Outcome: Cerebrospinal Fluid Changes - Interleukin 8 (IL8)
Description: IL-8 cytokine levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention.
Time Frame: at baseline and after 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 62.9 (5.27) | 102.5 (74.2)
  6 months | 91.6 (51.2) | 77.9 (19)

16. Secondary Outcome: Niacin Metabolite in Urine - Nicotinuric Acid NUA
Description: as for outcome 11
Time Frame: at baseline and after 6 months
Population: Plasma and urine samples will be tested to report levels of niacin and its metabolites. Higher value indicates higher niacin levels. A subset of the groups were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 23
ng/L
  at baseline | 3565.3 (7364.8) | 1021.8 (4538.7)
  6 months | 20132.9 (26789.4) | 2803.7 (8459.9)

17. Secondary Outcome: CSF Fluid Changes - Interleukin 1B (IL-1B)
Description: IL-1beta levels were tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention.
Time Frame: at baseline and 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  Baseline | 0.56 (0.8) | 0.28 (0.14)
  6 months | 0.21 (0.06) | 0.22 (0.07)

18. Secondary Outcome: Cerebrospinal Fluid (CSF) Changes - Macrophage Inflammatory Protein 1 Beta (MIP 1 Beta)
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of MIP-1 beta here.
Time Frame: at baseline and after 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pico grams per ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pico grams per ml
  baseline | 14.7 (5.02) | 9.3 (2.2)
  6 months | 15.9 (1.3) | 7.7 (4.2)

19. Secondary Outcome: Macrophage Changes
Description: The blood is tested to report G-protein coupled receptor 109A (GPR109A) levels in macrophages in M1 and M2 populations.
Time Frame: at baseline and after 6 months
Population: A subset of subjects were randomly selected for this measure and all the data is recorded here that was captured.
Measure: Mean (Standard Deviation); unit: percentage of macrophages
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 12 | 17
percentage of macrophages
  baseline | 54.08 (4.08) | 56 (4.5)
  6 months | 48.92 (3.9) | 54.5 (5.2)

20. Secondary Outcome: Niacin Metabolite Changes in Plasma - Nicotinamide (NAM)
Description: as for outcome 11
Time Frame: at baseline and after 6 months
Population: A subset of subjects were randomly selected for this analysis.
Measure: Mean (Standard Deviation); unit: uM/L
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 15 | 22
uM/L
  baseline | 0.43 (0.30) | 0.34 (0.19)
  6 months | 1.07 (0.46) | 0.38 (0.15)

21. Secondary Outcome: CSF Changes in Interferon Gamma (IF-gamma)
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of IF-gamma beta here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 0.21 (0.3) | 0.39 (0.39)
  6 months | 2.2 (2.3) | 0.89 (0.52)

22. Secondary Outcome: CSF Changes - Tumor Necrosis Factor - Alpha (TNF-alpha)
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of TNF-alpha here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 0.53 (0.87) | 0.18 (0.62)
  6 months | 0.23 (0.05) | 0.2 (0.31)

23. Secondary Outcome: Cerebral Spinal Fluid Changes - Interferon Gamma Induced Protein -10 (IP-10)
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of IP-10 here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 359.8 (193.5) | 512 (304.8)
  6 months | 936.2 (1018) | 514.5 (351.1)

24. Secondary Outcome: Cerebral Spinal Fluid (CSF) Changes - Monocyte Chemoattractant Protein 4 (MCP4)
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of MCP4 here.
Time Frame: at baseline and after 6 months
Population: Not all subjects donated CSF. All CSF samples are recorded here.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 24.6 (2.03) | 7.3 (8.1)
  6 months | 3.9 (5.6) | 6.7 (5.09)

25. Secondary Outcome: Cerebral Spinal Fluid (CSF) Changes - MIP1-alpha
Description: Inflammatory and non-inflammatory cytokines levels will be tested in cerebral spinal fluid (CSF) at baseline and 6 months after intervention. We are reporting levels of MIP1-alpha here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 3 | 10
pg/ml
  baseline | 17.8 (6) | 18.7 (3.8)
  6 months | 20.5 (18.2) | 17.3 (9.8)

26. Secondary Outcome: Plasma Cytokines - IF Gamma
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IF-gamma here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 16.2 (15.6) | 21 (33.1)
  6 months | 84.8 (287.7) | 15.95 (19.3)

27. Secondary Outcome: Plasma Cytokines - IL-10
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IL-10 here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 0.41 (0.28) | 0.41 (0.34)
  6 months | 0.5 (0.64) | 0.41 (0.28)

28. Secondary Outcome: Plasma Cytokines - IL1-B
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IL-1B here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 0.32 (0.34) | 0.37 (0.41)
  6 months | 0.23 (0.17) | 0.29 (0.28)

29. Secondary Outcome: Plasma Cytokines - IL-6
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IL-6 here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 5.7 (17.8) | 8.7 (34.2)
  6 months | 2.97 (4.25) | 11.04 (40.7)

30. Secondary Outcome: Plasma Cytokines - IL-8
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IL-8 here.
Time Frame: at baseline and after 6 Months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 6.7 (2.2) | 6.2 (2.1)
  6 months | 8.1 (3.5) | 6.6 (2.8)

31. Secondary Outcome: Plasma Cytokines - TNF-alpha
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of TNF-alpha here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 2.05 (4.7) | 0.96 (0.29)
  6 months | 2.26 (5.2) | 1.0 (0.31)

32. Secondary Outcome: Plasma Cytokines - IP-10
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of IP-10 here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 443.3 (197.3) | 402.7 (252.5)
  6 months | 542.1 (295.8) | 355.4 (158.6)

33. Secondary Outcome: Plasma Cytokines - MCP-4
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of MCP-4 here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 112.3 (73.8) | 104.6 (35.7)
  6 months | 106.4 (44) | 90.7 (41.3)

34. Secondary Outcome: Plasma Cytokines - MIP1-alpha
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of MIP1-alpha here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 23.3 (20.5) | 42.1 (116.7)
  6 months | 23.2 (9.3) | 38.9 (75.5)

35. Secondary Outcome: Plasma Cytokines - MIP1-beta
Description: Inflammatory and non-inflammatory cytokines levels will be tested in plasma at baseline and 6 months after intervention. We are reporting levels of MIP1-beta here.
Time Frame: at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 20 | 26
pg/ml
  baseline | 69.3 (26.1) | 65.8 (29.8)
  6 months | 65.5 (34.5) | 56 (24)

36. Secondary Outcome: Plasma Levels - Serotonin
Description: Plasma serotonin levels
Time Frame: at baseline and after 6 months
Population: a subset of the groups were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 16 | 14
mg/dL
  baseline | 84.2 (68.2) | 89.6 (60.5)
  6 months | 83 (75.2) | 64.2 (44.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Niacin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 7/21 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin (N=21) | Placebo (N=26)
flushing (Blood and lymphatic system disorders) | 7 (7) | 0 (0) — minimal flushing on either face or trunk

LIMITATIONS AND CAVEATS:
Additional studies are required including a larger cohort and multi-center to further generalize findings, as well as comparing niacin to placebo for longer than 6 months before optimal information can be obtained for use in clinical settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03462680/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT03462680/ICF_000.pdf